CLINICAL TRIAL: NCT01882361
Title: Opioid Relapse & HIV Risk: 48 Versus 24 Weeks of Injectable Extended Release Naltrexone
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 816019; R01DA033670 (NIH)
Record Dates: First submitted 2013-06-14; First posted 2013-06-20 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Opiate Dependence; Human Immunodeficiency Virus
Keywords: opioid addiction; opioid treatment; naloxone
MeSH Terms: conditions — Opioid-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — vivitrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- injectable naltrexone (Active Comparator): One dose of injectable extended release naltrexone (Vivitrol), 380mg dosage, given every four weeks in a 48-week trial.
  Interventions: Drug: injectable naltrexone
- placebo injection for naltrexone (Placebo Comparator): placebo comparator injection starting at week 24 in a 48-week trial.
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: injectable naltrexone — Vivitrol is an extended-release, microsphere formulation of naltrexone designed to be administered by intramuscular (IM) gluteal injection every 4 weeks or once a month. After IM injection, the naltrexone plasma concentration time profile is characterized by a transient initial peak, which occurs approximately 2 hours after injection, followed by a second peak observed approximately 2 - 3 days later. Beginning approximately 14 days after dosing, concentrations slowly decline, with measurable levels for greater than 1 month.
  Other Names: Vivitrol
  Arms: injectable naltrexone
Drug: placebo comparator — this placebo has no specific pharmacological activity
  Arms: placebo injection for naltrexone

SUMMARY:
To address the question of the comparison of two courses of Vivitrol with differing lengths in 130 HIV negative, consenting, opioid addicted patients who have completed inpatient treatment. Participants will be randomized under double blind conditions to a 24 or 48-week course of pharmacotherapy, along with bi-weekly drug counselling, over 48 weeks, with follow-ups at weeks 60 and 72. The 24-week cohort will receive Vivitrol placebo injections in weeks 24 to 48.

DETAILED DESCRIPTION:
1.2.1 Primary and Secondary Outcome Measures

Primary outcomes are:

1) Opiate positive urine tests; 2) HIV injecting risk.

Secondary outcomes are:

1) Time to relapse; 2) HIV sex risk; 3) Proportion of appointments kept; 6) Psychiatric symptoms; 7) Opioid craving; 8) Self-reported drug use; 9) Money spent for drugs; 10) Employment; 11) Arrests; 12) Overall adjustment; 12) Adverse events.

Hypotheses are that:

1. Primary outcomes will significantly favor the 48-week Vivitrol condition;
2. Five or more secondary outcomes will favor the 48-week condition; none will favor the 24-week condition.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative men and women 18 years of age or older who meet the Diagnostic and Statistical Manual of Mental Disorders 4th edition-Text Revision (DSM- IV-TR) criteria for opioid dependence
* Must be voluntarily seeking treatment for opioid dependence, with injection heroin as the drug and administration route of choice
* Must report sharing injection equipment during the past year
* Must have successfully completed inpatient detoxification at the Federal Medical Research Center for Psychiatry and Narcology (FMRCPN)
* Must have no current evidence of physiologic dependence
* Must have a stable address in Moscow with a telephone number where they can be reached
* If female, must have a negative pregnancy test and use of medically acceptable contraception if of childbearing age
* Must be able to provide informed consent as judged by the ability to read the consent and correctly answer 9 out of 10 questions about the study on a quiz

Exclusion Criteria:

* No current condition of psychosis (schizophrenia,paranoid disorder, mania)
* No history of major psychiatric disorders such as Schizophrenia, Major Depression with suicidal attempts, Bipolar I, uncontrolled epilepsy or other seizure disorder
* No current dependence (within the past year) to drugs other than prescription opiates or heroin, caffeine, marijuana, or nicotine based on the Diagnostic and Statistical Manual of Mental Disorders-Text Revision (DSM -IV-TR) criteria
* No current alcohol dependence or alcohol use disorder that would preclude successful completion of study procedures
* No current suicidal or homicidal ideation requiring immediate attention as determined at baseline assessment
* No cognitive impairment with inability to read and understand the consent
* No significant laboratory abnormality such as haemoglobin <10, hepatic transaminase levels >3 times upper limit of normal or serum creatinine that is >1.5 times upper limit of normal
* No legal charges with impending incarceration
* No concurrent participation in another treatment study
* Cannot be scheduled for surgery or be likely to require opioids for pain control in next 2 years
* Not currently taking naltrexone or currently receiving other treatment (pharmacological or behavioral) for drug dependence or currently receiving psychoactive medication
* Cannot have had receipt of any approved or investigational depot product administered into the gluteal muscle within 6 months before screening
* Cannot be on any excluded medication at screening or be anticipating the use of an excluded medication during the study period
* Cannot have participated in a clinical trial of a pharmacological agent within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Opiate positive urine tests | 12 months
  Reduction in drug use as seen by the primary urine outcomes will significantly favor the 48-week Vivitrol condition

SECONDARY OUTCOMES:
HIV sex risk | 12 months
  Participants will show significant HIV sex risk behaviors in the 48-week vivitrol condition.

OTHER OUTCOMES:
adverse events | 12 months
  No increase in known adverse events for the vivitrol arm as seen in other studies.

CONTACTS AND LOCATIONS:
Overall Officials: George E Woody, MD, Principal Investigator — University of Pennsylvania; Tatiana Klimenko, MD, PhD, Principal Investigator — Federal Medical Research Center for Psychiatry and Narcology (FMRC)
Locations (1):
- Federal Medical Research Center for Psychiatry and Narcology (FMRC), Moscow, Russia